CLINICAL TRIAL: NCT04412642
Title: Pilot Study to Assess the Feasibility of Self-administered Low Dose Methoxyflurane for Pain Relief During Minor Out-patient Urologic Procedures
Brief Title: Low Dose Methoxyflurane for Pain Relief During Minor Out-patient Urologic Procedures
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 431-2019
Record Dates: First submitted 2020-04-22; First posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-06

CONDITIONS: Pain, Acute
MeSH Terms: conditions — Acute Pain | interventions — Methoxyflurane

STUDY DESIGN:
Masking Description: no masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- methoxyflurane (Other): methoxyflurane
  Interventions: Drug: Methoxyflurane, MEOF

INTERVENTIONS:
Drug: Methoxyflurane, MEOF — As soon as possible following enrollment and initial procedures, the patient will be supplied with a PENTHROX™ kit which includes one inhaler containing 3 mL of MEOF for pain management. A member of the research team will train the patient to self-administer MEOF. PENTHROX™ is an approved (trademarked) product in Canada and is commercially available in a combination blister pack with one 3 mL sealed bottle and one PENTHROX™ inhaler with the Activated Carbon (AC) chamber.
  Other Names: Penthrox

SUMMARY:
The participant will be trained to self administer the drug and will be supplied with a PENTHROX commercial inhaler kit .The study nurse will train the participant and supervise its use during the procedure.Immediately following the procedure the participant will be asked to fill out two brief questionnaires. The study nurse will assess the participant for adverse event and will follow-up with a phone call 24 hours later.

DETAILED DESCRIPTION:
Many patients with chronic urological conditions require multiple and sometimes painful urological procedures. Ideally these procedures may be done in the cystoscopy suite without a general anesthetic. Low dose methoxyflurane, (MEOF)is a inhaled, self-administered non-opioid analgesic and has been approved by Health Canada's for the short-term relief of moderate to severe acute pain, associated with trauma or international medical procedures, in conscious adult patients. The brand name is PENTHROX.

This study is a single centre, pilot study to assess the feasibility of using a self-administrated, MEOF for pain relief during minor out-patient urological procedures. Eligible participants will receive a one time dose of the the study medication during a planned, outpatient urological procedure done under cystoscopy in the Cystoscopy clinic

ELIGIBILITY:
Inclusion Criteria:

1. Conscious adult patients >=
2. Patient is scheduled for cystoscopy And:

   * BOTOX injections for Overactive Bladder /Neuogenic Detrusor Overactivity,
   * Diagnostic hydrodistention for painful bladder syndrome
   * Biopsy or cauterization of bladder tumors
   * Biopsy, cauterization and/or injection of Hunner's lesions
   * Visual urethrotomy/bladder neck incision=/- injection of stricture
   * Evaluation of the complex urinary tract problems
3. Patient (patient/or patient's authorization legal representative) should understand the nature of the study and provide written informed consent
4. Patient is able to follow all study requirements and procedures and complete required questionnaires

Exclusion Criteria:

1. An altered level of consciousness, due to any cause, including head injury, drugs,or alcohol
2. Clinically significant renal impairment
3. Women of child bearing potential who are pregnant or peri partum, including labour
4. A history of liver dysfunction after previous MEOF use or other halogenated anesthetics
5. Hypersensitivity to MEOF or other halogenated anesthetics, or to butylated hydroxytoluene
6. Known or genetically susceptible to malignant hyperthermia or a history of severe adverse reactions in either patient or relatives
7. Exacerbation of an underlying condition (i.e., chronic pain)
8. Clinically evident or potential hemodynamic instability as per the opinion of the investigator
9. Clinically evident respiratory impairment as per the opinion of the investigator
10. Prior treatment with PENTHROX within 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-05-31 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction measured using the Patient Global assessment of Medication Performance (GMP)at the time of discharge | end of procedure
  Global assessment of Medication,which is an assessment, performed by the patient, of the patient's impression of how well the medication works. The patient is asked to rate the pain relief given by methoxyflurane using a 5-point likert scale - 0=poor;1=fair;2=good;3=very good;4=excellent

SECONDARY OUTCOMES:
The Overall/Maximum pain intensity experienced at any point during the procedure using a numeric rating scale | during the procedure
  Patient is asked to rate the intensity of the pain experienced using an 11-point numeric rating scale is used. A score of 0=no pain and a score of 10= worst pain possible
Percent patients requiring rescue medication | during the procedure
  Documentation of the use of rescue medication post administration of methooxyflurane Documenting first time of use of rescue medication, type of medication administered,dose and route
Safety outcome measure to assess percentage of patients requiring rescue medication | During the procedure;post procedure and at 24 hours post procedure (phone contact)
  Documentation of adverse events as safety outcome measure by the health care professional
Health professional impression of how well the medication worked measured using the Patient Global assessment of Medication Performance (GMP)at the time of discharge | end of procedure
  Global assessment of Medication Performance, is an assessment, performed by the health care professional, of their impression of how well the medication works. The health care professional is asked a single question "rate the pain relief provided by methoxyflurane using a 5-point likert scale - 0=poor;1=fair;2=good;3=very good;4=excellent
Assessment of how well the medication fulfilled the patient's expectations of pain relief using the Fulfillment of of Pain Relief Expectation Scale | end of procedure
  The patient is asked a single question "To what extent has your expectations regarding pain control been met?", using the Fulfillment of Pain Relief Expectation scale, which uses a 5-point Likert scale - 0=poor;1=fair;2=good;3=very good;4=excellent
Assessment of how well the medication fulfilled the health care professional's expectations of pain relief using the Fulfillment of of Pain Relief Expectation Scale | end of procedure
  The health care professional is asked a single question "To what extent has your expectations regarding pain control been met?", using the Fulfillment of Pain Relief Expectation scale, which uses a 5-point Likert scale - 0=poor;1=fair;2=good;3=very good;4=excellent

CONTACTS AND LOCATIONS:
Overall Officials: Sender Herschorn, MD, FRSC, Principal Investigator — Sunnybrook Health Sciences Centre